CLINICAL TRIAL: NCT07341815
Title: Efficacy of a Parental Support Intervention to Improve Communication of Advanced Cancer Patients With Adolescents and Young Adults
Brief Title: Parental Support Intervention in an Advanced Oncological Context
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Centre de Psycho-Oncologie (CPO) (Other); Jules Bordet Institute (Other); Erasme University Hospital (Other); Fonds Thierry Maricq & Véronique Detournay, Fondation Roi Baudouin, Belgium (Unknown); Association Jules Bordet (Unknown)
Responsible Party: Principal Investigator, Aurore Liénard, Pr, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE3373
Record Dates: First submitted 2025-12-16; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer; Cancer Recurrence; Hematological Cancer; Parent-Child Relations; Parenting; Communication
Keywords: Parental cancer; Parent-child communication; Parenting intervention; Advanced cancer; Adolescent Young Adult (AYA); Uncertainty
MeSH Terms: conditions — Neoplasm Metastasis; Communication

STUDY DESIGN:
Intervention Model Description: This study is a two-armed randomized trial with two groups receiving different interventions.
  In the "SOURCE - educational", patients benefit from a psycho-educational intervention based on an informational booklet. In the "SOURCE - experiential", the patients benefit from an intervention composed of a psycho-educational part (based on the same informational booklet) and a psycho-experiential intervention (role playing, relaxation exercises, etc.).
Masking Description: Participants are informed of the two existing intervention groups as soon as they are recruited. The participant and the assessor are blind during the first research interview (T1), since randomization is only given after the welcoming session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOURCE - educational (Active Comparator): Participants receive an informational brochure created for the study and take part in five or six intervention sessions lasting around 15 minutes each. These sessions focus on the informational content of the brochure, which is summarized in a PowerPoint presentation presented by the psycho-oncologist.
  Interventions: Device: Psycho-Education
- SOURCE - experiential (Experimental): Participants receive the same informational brochure and benefit from the same summary presentation in PowerPoint format as in the other arm. In addition, there is an experiential component, meaning that participants raise their specific questions/concerns related to the topics and work on them in a practical way with the psycho- oncologist.
  Interventions: Device: Psycho-Education; Behavioral: Psycho-Experiential

INTERVENTIONS:
Device: Psycho-Education — Supporting parents by providing useful informations and recommendations regarding communication with their children.
Behavioral: Psycho-Experiential — (1) Continuous support of parental self-efficacy about parental competence to communicate ; (2) Exercises about improving parental competence to communicate with their children (role-plays, transfer in the daily life).
  Arms: SOURCE - experiential

SUMMARY:
This prospective, two-arm randomized trial compares a psycho-educational program to a psycho-educational and experiential program for parents with advanced cancer. These two interventions aim to support parent-child communication about cancer, but we hypothesize that the combined intervention will be more effective for all studied communication variables.

DETAILED DESCRIPTION:
Background:

A recent review shows that 14-22% of patients with cancer are parents of underaged children or young adults. Following the cancer diagnosis, many parents report being concerned about the impact of the disease on their children and about how to communicate about the disease with them, especially about the uncertainty that is inherent in disease. In addition, they may report a decrease in their parental self-efficacy and in their parental skills to support their children. There are few randomized controlled trials designed to test the efficacy of parenting support interventions in oncology. Moreover, the existing studies use such varied designs and evaluation tools that there is no evidence-based practice in this area to date.

Methods:

The study is a prospective, two-armed randomized trial with two groups receiving either a psycho-educational program or a psycho-educational and experiential program.

This study is offered to patients with advanced cancer who have at least one child aged between 10 and 25 years. All participants must be interested in discussing how to communicate with their children about the disease.

All participants complete a baseline assessment (T1). Then, they are assigned randomly to one of the two intervention groups during a one-hour welcoming session. The second assessment interview (T2) is scheduled two weeks after the end of both interventions. The third assessment interview (T3) takes place 3 months after T2. Finally, a fourth short assessment (T4) is scheduled at the end of the current school year at T2. Moreover, participants are asked to complete a weekly assessment from T1 to T3 (during 6 months).

The "Supporting Open Uncertainty Responses and Communication Engagement : a psycho-educational program" (SOURCE - educational) and the "Supporting Open Uncertainty Responses and Communication Engagement : a psycho-educational and experiential program" (SOURCE - experiential) are based on an informational booklet designed to improve the knowledge of how to communicate with children, adolescents and young adults (AYAs), with a particular focus on communicating about the uncertainty inherent in disease. Both interventions are conducted in 5 to 6 manualized sessions by the same experienced psycho-oncologist.

In the "SOURCE - experiential", sessions last about 1,5 hour and are held in person or by teleconsultation. This intervention is based on support of parental self-efficacy and exercises about parental competence to communicate with their AYAs (role play and support of transfer in daily life).

In the "SOURCE - educational", sessions last about 15 minutes and are held by teleconsultation. It is a psycho-educational intervention aimed at supporting parents by providing information and recommendations regarding communication with AYAs and the potential impact of the disease on them.

Discussion:

It is hypothesized that the parental support provided in the psycho-educational and experiential program will be more effective than sessions offered in the context of the psycho-educational program for all the studied variables, even on communicating about uncertainty, a subject we know to be more sensitive.

EXPLORATORY PART OF THE STUDY Participants are also informed that, if they agree, their children aged between 10 and 25 will be invited to participate to an exploratory part of the study. To be eligible to participate in this exploratory part, AYAs must have a strong command of French, and be aware that their parent has a disease (whether or not called "cancer") and that their parent receive or has received a treatment for that disease. AYAs are excluded if they are living completely independently, if they have severe neurological or psychiatric disorders, or if they are in special-needs education. In order to participate, AYAs must sign a consent document. If they are minors, an additional consent document must be signed by their ill parent, and the co-parent must give an oral consent.A non-participation of the AYA to the study does not affect the inclusion of their parent in the study.

Exploratory outcomes are: (1) communication about cancer or its consequences in the family from the AYA's perspective, (2) AYA's communication wishes, (3) future expectations of parental disease and treatments and (4) global quality of life. Questionnaires are completed three times, at most 48 hours apart from the T1, T2, and T3 of their parent.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer, recurrence of cancer or certain types of hematological cancer (chronic disease, acute leukemia, multiple myeloma or lymphoma recurrence)
* Have at least one child aged between 10 and 25 years
* Wish to benefit from a psychological intervention about communication with their children about cancer or its consequences
* Able to read and speak French
* Accept to give their written informed consent

Exclusion Criteria:

* Severe neurological disorder
* Severe psychiatric disorder
* (Pre-)terminal phase of cancer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of parental communication with their children about cancer or its consequences | Weeks 2 to 26 (weekly assessment).
  In the weekly assessment, participants are asked how many moments of communication they had with their child(ren) about cancer, treatments, or their consequences during the past week. This item measures the frequency of communication.
Quality of parental communication with their children about cancer or its consequences | Weeks 2 to 26 (weekly assessment).
  A composite communication quality score will be computed for each communication moment reported in the weekly assessments. The score will be based on several dimensions:
  1. Initiative, indicating whether the communication was initiated by the parent (yes/no);
  2. Duration of the communication moment, reported in minutes;
  3. Parental self-efficacy, defined as the perceived ability to inform, listen, answer questions, and reassure, each rated on a 0-10 Likert scale (0 = not at all capable; 10 = completely capable);
  4. Comfort during the communication, assessed separately for the parent and the child using a 0-10 Likert scale (0 = not at all comfortable; 10 = extremely comfortable);
  5. Disease-related topics discussed (yes/no);
  6. Emotional expression, assessed using two yes/no items indicating whether the parent expressed their emotional experience and/or addressed the child's emotional experience related to the disease.
  Higher scores reflect better communication quality.
Parental communication difficulties | Baseline (T1), week 12 (T2) and week 26 (T3).
  The level of perceived difficulties to communicate is assessed through one item 10-point Likert scale (0 = not at all certain; 10 = absolutely certain).
Parental self-efficacy regarding the communication with their children about cancer or its consequences | Baseline (T1), week 12 (T2) and week 26 (T3).
  The level of self-efficacy to communicate is assessed through 27 items covering a list of disease-related communication topics (3 subscales of 9 items each : "I know how to communicate", "I am able to communicate" and "I am comfortable to communicate") 10-point Likert scale (0 = not at all certain; 10 = absolutely certain).
  The total score is obtained by summing the responses to all 27 items (maximum score = 270), and subscale scores are calculated by summing the 9 corresponding items (maximum score = 90).
Participants' communication behaviors | Baseline (T1), week 12 (T2) and week 26 (T3).
  The participants' communication behaviors about cancer are assessed through a 13 items 4- point Likert scale (0 = no; 1 = rather no; 2 = rather yes; 3 = yes).
  Items are phrased as statements such as "I talked about…" and cover a range of disease-related topics. A total score of disease-related communication repertoire is calculated by summing the responses to all items, with higher scores indicating a broader range of topics addressed.
Theoretical knowledge about the cancer-related concerns of children of different ages | Baseline (T1), week 12 (T2) and week 26 (T3).
  The level of theoretical knowledge about children's concerns about cancer is assessed through a true-false questionnaire containing 12 items.
  Correct answers were previously determined by experts in the field. Each correct response is scored as 1 point, and each incorrect response as 0 point. A total knowledge score is obtained by summing the scores across all items, with higher scores reflecting greater theoretical knowledge.
Under- / Over- communication | Baseline (T1), week 12 (T2) and week 26 (T3).
  Over- and under-communication are assessed using 10 items, divided into two subscales of 5 items each, rated on a 10-point Likert scale (0 = not at all certain; 10 = absolutely certain). Each subscale score ranges from 0 to 50.
  For the total score, the under-communication subscale is assigned negative values and the over-communication subscale positive values; the two are then summed, resulting in a possible range from -50 to +50. Higher positive scores indicate a stronger tendency toward over-communication, whereas lower (negative) scores indicate a stronger tendency toward under-communication about cancer.
Parental perception of their children's experience of cancer | Baseline (T1), week 12 (T2) and week 26 (T3).
  The parental perception of their children's experience of cancer is assessed through 8 items rated on a 10-point Likert scale (0 = not at all certain; 10 = absolutely certain). A higher item score indicates that the parent feels they have a good understanding of their children's experience regarding the disease-related topic.
  The total score, which can range from 0 to 80, reflects the parent's overall perception of their children's experience of the disease.

SECONDARY OUTCOMES:
Perceived children's communication behaviors | Baseline (T1), week 12 (T2) and week 26 (T3).
  Perceived children's communication behaviors are assessed through a 12-item, 4-point Likert scale (0 = no; 1 = rather no; 2 = rather yes; 3 = yes). This questionnaire explores disease-related topics the child spontaneously brought up during conversations. The total score, obtained by summing the responses to all items, reflects the breadth of the child's spontaneous communication repertoire regarding the disease.
Parental self-efficacy in general | Baseline (T1), week 12 (T2) and week 26 (T3).
  The level of parental self-efficacy in general is assessed through one validated item (Moore et al., 2015) rated on a 10-point Likert scale (0 = not at all certain; 10 = absolutely certain).
Children's academic performance | Baseline (T1), at the end of the current academic year at the time of week 12 (T4).
  The authors developed a questionnaire to assess the academic performance of participants' children. This questionnaire explores the child's current level of education (i.e., current school grade if the child is still enrolled), as well as retrospective information about the previous school year, including the jury's decision (pass with or without conditions, or failure), the child's overall grade point average, and the number of subjects in which the child failed. Additionally, the questionnaire collects information on the total number of grade retentions since the beginning of the child's schooling.
Participant's perception of their AYA's global quality of life (KIDSCREEN) | Baseline (T1), week 12 (T2) and week 26 (T3).
  Children's global quality of life is assessed using the KIDSCREEN questionnaire. The KIDSCREEN is available in both self-reported and hetero-reported versions; the latter is used to gather parents' perspectives on their children's quality of life. We used a 36-item version, rated on a 5-point Likert scale (with response options varying across items).
  In addition to a total score-calculated by summing responses across all 36 items-the questionnaire provides results on seven subscales: (1) Physical activities and health (5 items), (2) Child's feelings (3 items), (3) General mood (7 items), (4) Child's free time (4 items), (5) At home (6 items), (6) Friends (5 items), and (7) At school/university (6 items). For the last subscale, a "not applicable" option is available if the child is no longer enrolled in school.
Parents' Distress associated with parenting | Baseline (T1), week 12 (T2) and week 26 (T3).
  Parenting concerns related to cancer are assessed through the PCQ (Parenting Concerns Questionnaire). This questionnaire contains 14 items 5-point Likert scale (1 = not at all concerned; 5 = extremely concerned). The subscales of the PCQ are: "practical impact of illness on child", "emotional impact of illness on child" and "concerns about coparent". However, the third PCQ subscale has been adapted to measure concerns in relation to the entourage as a whole.
Expectations and Benefits of the intervention | Baseline (T1), week 12 (T2).
  The BENEVAL is a tool used in T1 to assess participants' expectations of the intervention and in T2 to assess participants' perceived benefits (Razavi, Wauthia, Bodart, & Servais, 2014). It contains 11 domains, each with sub-questions (between 2 and 9 sub-questions) to be answered on a 5-point Lickert scale (from not at all to very much).
Perceived usefulness of the interventions | Week 12 (T2).
  Perceived usefulness of the interventions is assessed using a 10-item, 10-point Likert scale (0 = not at all certain; 10 = absolutely certain). A total score is calculated by summing the responses across all items.

OTHER OUTCOMES:
Communication about cancer or its consequences in the family from the AYA perspective | Baseline (T1), week 12 (T2) and week 26 (T3).
  Communication about cancer or its consequences in the family from the AYA perspective is assessed through 10 items 10-point Likert scale (0 = not at all true; 10 = absolutely true).
AYA's communication wishes | Baseline (T1), week 12 (T2) and week 26 (T3).
  AYA communication wishes are assessed through 10 items 10-point Likert scale (0 = not at all true; 10 = absolutely true).
AYA's future expectations of parental disease and treatments | Baseline (T1), week 12 (T2) and week 26 (T3).
  AYA's future expectations regarding parental disease and treatments are assessed using a 10-item measure. For each item, participants are asked to (1) choose between two proposed outcomes for a given situation-one optimistic and one pessimistic-and (2) indicate their level of certainty that this outcome will occur, selecting from three options: might, probably, or definitely.
  Among the 10 situations presented, 6 are neutral and realistic, while 4 are specifically related to the disease.
  Scoring is based on both the valence of the choice and the level of certainty. If the optimistic outcome is chosen, the score is assigned a positive sign; if the pessimistic outcome is chosen, the score is negative. The level of certainty determines the absolute value of the score: might = 1, probably = 2, and definitely = 3.
  Scores are summed separately for the two subscales.
Participant's future expectations of disease and treatments | Baseline (T1), week 12 (T2) and week 26 (T3).
  This questionnaire should only be completed by the parent if one of his or her children is participating in the study. Participant's future expectations of disease and treatments are assessed using a 10-item measure. For each item, participants are asked to (1) choose between two proposed outcomes for a given situation-one optimistic and one pessimistic - and (2) indicate their level of certainty that this outcome will occur, selecting from three options : might, probably, or definitely.
  Among the 10 situations presented, 6 are neutral and realistic, while 4 are specifically related to the disease.
  Scoring is based on both the valence of the choice and the level of certainty. If the optimistic outcome is chosen, the score is assigned a positive sign; if the pessimistic outcome is chosen, the score is negative. The level of certainty determines the absolute value of the score: might = 1, probably = 2, and definitely = 3.
  Scores are summed separately for the two subscales.
AYA's perception of their own global quality of life (KIDSCREEN) | Baseline (T1), week 12 (T2) and week 26 (T3).
  AYA global quality of life is assessed through the KIDSCREEN. The KIDSCREEN is available in a self-reported or hetero-reported version. The AYAs complete the self-reported version. We used 36 items 5-point Likert scale (the positions on the scale change from one item to another).
  In addition to a total score-calculated by summing responses across all 36 items-the questionnaire provides results on seven subscales: (1) Physical activities and health (5 items), (2) Feelings (3 items), (3) General mood (7 items), (4) Free time (4 items), (5) At home (6 items), (6) Friends (5 items), and (7) At school/university (6 items). For the last subscale, a "not applicable" option is available if the child is no longer enrolled in school.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: Undecided